CLINICAL TRIAL: NCT00040573
Title: A Phase I/II Open Label, Single Dose Study of Intracavitary Administered 131I-TM-601 in Adult Patients With Recurrent High-Grade Glioma.
Brief Title: Safety and Tolerability Study of 131I-TM-601 to Treat Adult Patients With Recurrent Glioma.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: TransMolecular (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TM601-001
Record Dates: First submitted 2002-06-29; First posted 2002-07-02 (Estimated); Last update posted 2009-03-31 (Estimated); Status verified 2009-03

CONDITIONS: Glioma; Brain Neoplasm
Keywords: Brain neoplasm; Clinical trial, phase I/II
MeSH Terms: conditions — Glioma; Brain Neoplasms | interventions — Chlorotoxin

INTERVENTIONS:
Drug: 131I-TM-601

SUMMARY:
This drug is being developed to treat a type of brain cancer, glioma. This study was designed to determine a safe and well tolerated dose. Patients must have had prior treatment for their glioma and be eligible for removal of their recurring tumor.

DETAILED DESCRIPTION:
This is an open label single-dose study to be conducted in 18 evaluable patients with recurrent high-grade glioma. Patient will undergone debulking surgery and ventricular access device placement into the tumor cavity for administration of 131I-TM-601. High-grade glioma includes glioblastoma multiforme, anaplastic astrocytoma, anaplastic oligo-astrocytoma and gliosarcoma. The amount of 131I will remain constant. Three doses of TM-601 will be administered using a dose escalating scheme.

ELIGIBILITY:
* Patient must have given informed consent
* Patient must have histologically confirmed supratentorial malignant glioma
* Patients must have recovered from toxicity of prior therapy
* Patients must be eligble for resection of the recurrent tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18
Dates: Start 2002-06; Study Completion 2003-08

CONTACTS AND LOCATIONS:
Overall Officials: Diana M Hablitz, MSNCRNP, Study Director — TransMolecular
Locations (3):
- United States (3):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City of Hope, Duarte, California
  - Saint Louis University, St Louis, Missouri